CLINICAL TRIAL: NCT03183349
Title: Immediate Implant Placement With Platlet Rich Fibrin as Space Filling Material Versus the Use of Deprotienized Bovine Bone (Tutogen) in Maxillary Premolars. A Randomized Controlled Clinical Trial
Brief Title: Immediate Implant Placement With Platlet Rich Fibrin as Space Filling Material Versus the Use of Deprotienized Bovine Bone (Tutogen) in Maxillary Premolars.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed mohamed awad elbrashy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cebc.Cairouni
Record Dates: First submitted 2017-06-06; First posted 2017-06-12 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Immediate Dental Implant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet rich fibrin (Experimental): immediate implant grafting
  Interventions: Procedure: deprotienized bovine bone (tutogen)
- deprotienized bovine bone (tutogen) (Active Comparator): immediate implant grafting
  Interventions: Procedure: platelet rich fibrin

INTERVENTIONS:
Procedure: deprotienized bovine bone (tutogen)
  Arms: platelet rich fibrin
Procedure: platelet rich fibrin
  Arms: deprotienized bovine bone (tutogen)

SUMMARY:
20 subjects suffering from non restorable maxillary premolar teeth will be randomly devided into two groups. the selected teeth will be extracted and immeiate implants will be placed in all subjects. the first group will recieve deprotienized bovine bone (tutogen) to fill the buccal space between the implant and the bone, the second group will recieve platlet rich fibrin to fill the buccal space between the implant and the bone

ELIGIBILITY:
Inclusion Criteria:

* non restorable maxillary premolars non smoker free from any systemic disease or medication that could impair normal bone healing

Exclusion Criteria:

* any systemic disease that could affect bone healing patient with lesion related to the surgical site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Patient morbidity | 14 days
  patient pain level on pain scale using pain chart

SECONDARY OUTCOMES:
crestal bone loss | 3 months
  radiographic analysis computing amount of crestal bone loss around implants using cone beam computed tomography
implants stability quotient | 3 months
  implant stability measured using resonance frequency analysis

IPD SHARING:
Plan to Share IPD: Yes